CLINICAL TRIAL: NCT02676375
Title: Nicotine Receptor Density & Response to Nicotine Patch: Pt 2 Extended Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brentwood Biomedical Research Institute (Other)
Responsible Party: Principal Investigator, Arthur Brody, Research Psychiatrist, Brentwood Biomedical Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0024
Record Dates: First submitted 2016-02-04; First posted 2016-02-08 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Smoking Cessation; Schizophrenia
MeSH Terms: conditions — Smoking Cessation; Schizophrenia | interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Monotherapy (Other): Treatment as usual starting with one smoking cessation medication plus group therapy.
  Interventions: Drug: Monotherapy
- Combination Extended Treatment (Experimental): Extended treatment with multiple standard medications plus group therapy.
  Interventions: Drug: Combination Bupropion + NRTs; Other: Extended Treatment
- Combination Extended Treatment + Home Visits/Calls (Experimental): Extended treatment with multiple standard medications plus group therapy plus home visits.
  Interventions: Drug: Combination Bupropion + NRTs; Other: Extended Treatment; Other: Home Visits & Calls

INTERVENTIONS:
Drug: Combination Bupropion + NRTs
  Arms: Combination Extended Treatment; Combination Extended Treatment + Home Visits/Calls
Other: Extended Treatment
  Arms: Combination Extended Treatment; Combination Extended Treatment + Home Visits/Calls
Other: Home Visits & Calls
  Arms: Combination Extended Treatment + Home Visits/Calls
Drug: Monotherapy
  Arms: Standard Monotherapy

SUMMARY:
The study investigators will enroll 45 treatment seeking, cigarette smokers with a Diagnostic and Statistical Manual (DSM-IV) diagnosis of schizophrenia who will be randomly assigned into three arms of treatment for smoking cessation treatment, receiving either 1. Control: "standard therapy" (n=15), including stepwise monotherapy of nicotine patch or bupropion sustained release, 2. Extended treatment with combination bupropion, nicotine patch, and nicotine lozenge for 6 months (n=15), or 3. Extended treatment with combination bupropion, nicotine patch, and nicotine lozenge for 6 months with home visits (n=15) and phone calls to the home or living facility. During all treatments, participants will receive weekly smoking cessation group counseling, as is standard for smoking cessation treatment. At the time of enrollment, participants will complete a one-study visit lead-in to complete baseline assessments, psychological and medical evaluation, and comprehensive assessment of drug use to determine study eligibility. Once determined to be eligible for the trial, participants will be randomly assigned to one of the treatment arms using a randomization procedure. The "standard therapy" treatment arm, or control group, will receive either nicotine patch taper starting at 21 milligrams (mg) daily, nicotine lozenge as needed, and/or bupropion sustained release at 150mg daily for 3 days, then 150 mg twice a day for a total of 12 weeks. The extended therapy arm will start the nicotine patch at 21mg daily with as needed nicotine lozenge for breakthrough cravings and initiation of bupropion sustained release at 150mg daily for 3 days a week prior to starting nicotine replacement, then 150 mg twice daily for 6 months (as tolerated). The third arm will be identical to the second arm except for the added home visit intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans 21 years of age or older;
2. meet DSM-IV criteria for Schizophrenia or Schizoaffective disorder based on clinical interview
3. meet DSM-IV criteria for nicotine dependence
4. must report smoking >10 cigarettes daily and positive CO exhalation >8ppm
5. seeking treatment for nicotine dependence;
6. willing and able to comply with study procedures;
7. willing and able to provide written informed consent;
8. if female, not pregnant or lactating and willing to use a medically reliable method of birth control during the trial (e.g., birth control pills, Depo-Provera, and/or condoms with spermicide).
9. Must be clinically stable (i.e., no inpatient hospitalizations for 3 months prior to enrollment, no changes in medication in the four weeks prior to enrollment)

Exclusion Criteria:

1. current or past history of cardiovascular disease including myocardial infarction, acute coronary syndrome, angina pectoris, coronary artery disease, atrial fibrillation/flutter, cor pulmonale, arrhythmia other than sinus tachycardia or sinus bradycardia, or an EKG suggesting any of these;
2. systolic blood pressure greater than 160 or diastolic blood pressure greater than 100 (i.e. cutoffs for stage 2 hypertension)
3. a history of angioedema;
4. renal impairment (CrCl < 50);
5. a current neurological disorder (e.g., organic brain disease, dementia) or a medical history which would make study agent compliance difficult or which would compromise informed consent;
6. a history of attempted suicide (lifetime) and/or suicidal ideation in the past year as assessed by the C-SSRS;
7. currently on prescription medication that is contraindicated for use with bupropion;
8. currently using any form of nicotine replacement therapy;
9. current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV within the past 6 months;
10. a history of sensitivity to bupropion or nicotine replacement;
11. any history of seizures or seizure disorder;
12. a history of serious head injury (ie, loss of consciousness longer than 1 hour, no neuropsychological sequelae, no cognitive rehabilitation treatment post head injury
13. evidence of substance or alcohol dependence in the past six months; evidence of substance or alcohol abuse in the past month;
14. sedatives or benzodiazepine use within 12 hours of testing based on urine toxicology screening
15. history of mental retardation or developmental disability based on chart review
16. psychiatric hospitalization during study participation
17. history of an eating disorder
18. have a medical condition that could be made worse by treatment with nicotine, including poorly controlled insulin dependent diabetes, uncontrolled hyperthyroidism, pheochromocytoma, severe oropharyngeal, esophageal, or peptic ulcer disease, or severe renal or hepatic impairment as determined via the baseline medical history and physical exam
19. have an allergy to adhesive tape or latex or serious dermatologic disease (excluding minor skin conditions such as mild eczema) due to potential for skin allergy to patch
20. have a known allergy to nicotine or any component of the nicotine patches
21. be pregnant or sexually active and not using reliable birth control methods consistently (for females)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- West Los Angeles Veterans Affairs Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Monotherapy: Treatment as usual starting with one smoking cessation medication plus group therapy.
  Monotherapy
- Combination Extended Treatment: Extended treatment with multiple standard medications plus group therapy.
  Combination Bupropion + NRTs
  Extended Treatment
- Combination Extended Treatment + Home Visits/Calls: Extended treatment with multiple standard medications plus group therapy plus home visits.
  Combination Bupropion + NRTs
  Extended Treatment
  Home Visits & Calls
Period: Overall Study
Arm/Group | Standard Monotherapy | Combination Extended Treatment | Combination Extended Treatment + Home Visits/Calls
Started | 14 | 14 | 14
Completed | 13 | 10 | 11
Not Completed | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Monotherapy | Combination Extended Treatment | Combination Extended Treatment + Home Visits/Calls | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (8) | 56 (10) | 56 (8) | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 14 | 14 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Carbon Monoxide (CO) as Parts Per Million (PPM)
Description: Weekly measurements of expired carbon monoxide in the units of parts per million (PPM) participants to evaluate abstinence from smoking (a value equal to or less than 3 PPM is considered abstinent).
Time Frame: Measured week 0, 12, and 26
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Standard Monotherapy | Combination Extended Treatment | Combination Extended Treatment + Home Visits/Calls
Number analyzed (Participants) | 13 | 10 | 11
ppm
  Week 0 | 11.5 (5.1) | 12.3 (9.9) | 12.0 (4.8)
  Week 12 | 7.8 (7.9) | 5.6 (4.5) | 5.9 (4.5)
  Week 26 | 10.7 (7.6) | 5.0 (3.3) | 5.0 (4.4)

ADVERSE EVENTS:
Time Frame: For the 26 weeks the study was conducted.
Description: Due to the nature of the study, there was not a substantial risk for serious adverse events or mortality. Non serious adverse events were recorded non systematically.
Arm/Group | Standard Monotherapy | Combination Extended Treatment | Combination Extended Treatment + Home Visits/Calls
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 6/13 | 3/10 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Monotherapy (N=13) | Combination Extended Treatment (N=10) | Combination Extended Treatment + Home Visits/Calls (N=11)
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Vivid dreams (Psychiatric disorders) | 1 | 2 | 0
Rash (with the patch) (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Modest sample size lacked power to differentiate between the COMB-EXT groups with/without HV; no control group other than TAU; no motivation to quit rating scale; no biochemical (plasma, salivary, urine) measures taken to ensure abstinence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No